CLINICAL TRIAL: NCT02224404
Title: Open, Non-comparative, Multi-centre Post Market Clinical Follow-up Investigation to Evaluate Performance and Safety on Pressure Ulcers, PU, When Using Exufiber as Intended
Brief Title: Post Market Clinical Follow-up Investigation to Evaluate Performance and Safety on Pressure Ulcers, PU, When Using Exufiber as Intended
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEXU02
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2014-08

CONDITIONS: Pressure Ulcers
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fast Gelling Dressing (Experimental)
  Interventions: Device: Fast Gelling Dressing (Exufiber)

INTERVENTIONS:
Device: Fast Gelling Dressing (Exufiber)

SUMMARY:
The primary objective of this post market clinical follow-up (PMCF) investigation is to evaluate performance and safety of Exufiber when used as intended in Stage II-IV pressure ulcers (PU).

ELIGIBILITY:
Inclusion Criteria:

1. Both gender ≥18 years old.
2. Subjects with Stage 2, 3 or 4 cavity pressure ulcer (acc to EPUAP)
3. Exuding pressure ulcer
4. Signed Informed Consent.

Exclusion Criteria:

1. Known allergy/hypersensitivity to the dressing.
2. Infected wounds, (2 signs of infection/local inflammation and a positive swab)
3. Stage 1 PU
4. Dry wounds
5. Subjects who will have problems following the protocol
6. Subjects included in other ongoing clinical investigation at present or during the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Beele, prof. dr, Principal Investigator — University Hospital Gent, Belgium
Locations (4):
- Belgium (3):
  - Dermatologie Campus Kennedylaan, Kortrijk, Kortrijk
  - Dep. of Plastic Surgery UZ Bruzzel, Brussels
  - University Hospital Gent, Belgium, Ghent
- Töölö Hospital, Helsinki, Finland

RESULTS

PARTICIPANT FLOW:
Groups:
- Fast Gelling Dressing: Fast Gelling Dressing (Exufiber)
Period: Overall Study
Arm/Group | Fast Gelling Dressing
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fast Gelling Dressing
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (19.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 7
Region of Enrollment [Number; unit: participants]
  Belgium | 14
  Finland | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Worsening in Peri-Skin Wound.(Maceration From Baseline to 6 Weeks)
Description: the subjects will be measured by the following variables; maceration,
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Fast Gelling Dressing
Number analyzed (Participants) | 21
participants | 2

2. Secondary Outcome: Evaluate the Level of Pain at Week 6 Changes in Wound Status, Clinician's and Subject's Opinion, and Technical Performance
Description: Pain during product removal at week 6, measured by Visual Analog scale.This will be measured by the following variables; visual analog scale, 0=no pain, 100= worst pain, scale from 0-100 mm
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Fast Gelling Dressing
Number analyzed (Participants) | 21
units on a scale | 0 [0 to 50]

ADVERSE EVENTS:
Arm/Group | Fast Gelling Dressing
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 1/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fast Gelling Dressing (N=21)
Nausea and vomiting (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fast Gelling Dressing (N=21)
Periwound redness (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less